CLINICAL TRIAL: NCT00807989
Title: An Open Label, Randomized, Multicenter Clinical Trial to Compare the Efficacy and Safety of Lamotrigine / Valproate Coadministration and Carbamazepine as Initial Pharmacotherapy in Epilepsies (Phase Ⅳ)
Brief Title: The Efficacy and Safety of Low Dose Combination of LTG and VPA Compared to CBZ Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109887
Record Dates: First submitted 2008-11-28; First posted 2008-12-15 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Carbamazepine; Lamotrigine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbamazepine (Active Comparator): Carbamazepine
  Interventions: Drug: Carbamazepine
- Lamotrigine/Valproate (Experimental): Lamotrigine and Valproate combination therapy
  Interventions: Drug: Lamotrigine/Valproate

INTERVENTIONS:
Drug: Carbamazepine
  Arms: Carbamazepine
Drug: Lamotrigine/Valproate
  Arms: Lamotrigine/Valproate

SUMMARY:
To evaluate the efficacy of usual monotherapy and low dose combination of Lamotrigine and Valproate. Low dose combination may be more effective and tolerable because they are low dose and VPA reduce Lamotrigine metabolism.

DETAILED DESCRIPTION:
An Open label, Randomized, Multicenter Clinical Trial to Compare the Efficacy and Safety of Lamotrigine / Valproate Coadministration and Carbamazepine as Initial Pharmacotherapy in Epilepsies

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16yr old
* Who are diagnosed as epilepsy definitely
* Who have minimum 2 unprovoked seizures and minimum 1 seizure in previous 3 months
* Who need AED therapy and no AED medication for previous 1 year (exclude emergency medication for less than 2weeks)
* Who is not pregnant
* Who can report seizure diary by him/herself or caregiver
* Who agree to this trial and provide informed consent.
* Type of seizures : of generalized tonic-clonic, complex partial, and/or simple partial motor seizures;

Exclusion Criteria:

* Who has progressive CNS disease.
* Has serious systemic or psychiatric disease
* Who is not suitable by investigator(uncooperative)
* Who can not fill up diary check card
* Is pregnant, breastfeeding, or planning to become pregnant
* Exclusion - absence s. juvenile myoclonic epilepsy, atonic seizure, alcohol or other substance abusers, mental retardation etc.
* Who cancels to agree to this trial and provide informed consent.
* ALT, AST, bilirubin and BUN/Cr levels are more than twice normal range of them
* WBC value is 2000 and less, Hb value is 9.0 and less, platelet count is 100,000 and less in CBC
* Who took investigation products before participating this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung-In Lee, Principal Investigator — Yonsei Univ.; Kyoung Heo, Principal Investigator — Yonsei Univ.; Sang-Kun Lee, Principal Investigator — Seoul National Univ.; Sang-Ahm Lee, Principal Investigator — Ulsan Univ.; Dong-Jin Shin, Principal Investigator — Gacheon Univ.; Hong-Ki Song, Principal Investigator — Hallym Univ.; Young-In Kim, Principal Investigator — Catholic Univ.; Se-Jin Lee, Principal Investigator — Youngnam Univ.; Sang-Ho Kim, Principal Investigator — Donga Univ.; Myung-Gyu Kim, Principal Investigator — Cheonnam Univ.; Yo-Sik Kim, Principal Investigator — Wonkwang Univ.; Sang-Do Lee, Principal Investigator — Dongsan Hosp.; Sung-Eun Kim, Principal Investigator — Pusan-Bak Hosp.; Sung-Pa Park, Principal Investigator — Kyungbuk Univ.; Joo-Yong Kim, Principal Investigator — Hanrim Univ.; Ok-Jun Kim, Principal Investigator — Bundang Cha; Soon-Ki Noh, Principal Investigator — Bong-Sang Hosp.; Hyang-Woon Lee, Principal Investigator — I-wha Univ.; Jae-Moon Kim, Principal Investigator — Chungnam Univ.
Locations (1):
- Yonsei Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbamazepine: Carbamazepine 100mg/day for the first two weeks. At next two weeks, dose of Carbamazepine was increased to 200mg/day in two divided doses
- Lamotrigine/Valproate: Lamotrigine and Valproate combination therapy
  Lamotrigine 25mg/day for the first two weeks. At next two weeks, LTG 50 mg once a day
Period: Overall Study
Arm/Group | Carbamazepine | Lamotrigine/Valproate
Started | 107 | 100
Completed | 104 | 98
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine/Valproate: Lamotrigine and Valproate combination therapy
  Lamotrigine/Valproate
- Total: Total of all reporting groups
Arm/Group | Carbamazepine | Lamotrigine/Valproate | Total
Number analyzed (Participants) | 104 | 98 | 202
Age, Continuous [Mean (Standard Deviation); unit: Year] | 33.2 (14.6) | 36.5 (13.7) | 34.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 53 | 50 | 103
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 104 | 98 | 202

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate After 52 Weeks Maintenance Period
Description: * Retention rate means completion rate (CR), the proportion of patients who have completed the 60-week study as planned.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Carbamazepine | Lamotrigine/Valproate
Number analyzed (Participants) | 104 | 98
participants | 104 | 98

2. Secondary Outcome: Seizure Free Rate for 24 Weeks at Initial Target Dose
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Carbamazepine | Lamotrigine/Valproate
Number analyzed (Participants) | 90 | 78
participants | 51 | 59

3. Secondary Outcome: Seizure Free Rate for 52 Weeks at Initial Target Dose
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Carbamazepine | Lamotrigine/Valproate
Number analyzed (Participants) | 90 | 78
participants | 43 | 50

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Carbamazepine | Lamotrigine/Valproate
Serious Adverse Events (participants affected / at risk) | 9/104 | 0/98
Other Adverse Events (participants affected / at risk) | 60/104 | 59/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbamazepine (N=104) | Lamotrigine/Valproate (N=98)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Atonic seizures (Nervous system disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbamazepine (N=104) | Lamotrigine/Valproate (N=98)
Headache (Nervous system disorders) | 26 (29) | 26 (52)
Dizziness (Nervous system disorders) | 18 (23) | 17 (18)
Somnolence (Nervous system disorders) | 14 (15) | 12 (12)
Memory impairment (Nervous system disorders) | 10 (14) | 5 (5)
Tremor (Nervous system disorders) | 2 (2) | 11 (11)
Skin rash (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 5 (7)
Weight gain (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Nasopharyngitis (Infections and infestations) | 7 (9) | 10 (26)
Fatigue (General disorders) | 10 (10) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days